CLINICAL TRIAL: NCT02106884
Title: Randomized Crossover Trial to Assess the Effects and Quality of Life in Patients With Locally Advanced or Metastatic Pancreatic Cancer Treated With Gemcitabine in Combination With Nab-paclitaxel: QOLINPAC
Brief Title: Quality of Life in Locally Advanced or Metastatic Pancreatic Cancer Treated With Gemcitabine and Nab-paclitaxel
Acronym: QOLINPAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s56122; 2013-004101-75 (EudraCT Number); AX-CL-PANC-PI-003568 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2014-01-21; First posted 2014-04-08 (Estimated); Results first posted 2019-10-24 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Locally advanced; Metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Nab-paclitaxel - IV - 125 mg/m2 - 3xq4wks Gemcitabine - IV - 1000 mg/m2 - 3xq4wks
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine
- Arm B (Active Comparator): Gemcitabine - IV - 1000 mg/m2 - 3xq4wks
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Nab-paclitaxel
  Other Names: Abraxane, EU/1/07/428/001, L01CD01
  Arms: Arm A
Drug: Gemcitabine
  Other Names: Gemzar

SUMMARY:
This was a quality of life (QOL) study done in the context of a randomized trial in locally advanced or metastatic pancreatic cancer. Eligible patients were randomized to receive either the combination of nab-paclitaxel/gemcitabine or standard gemcitabine monotherapy. The combination regimen of nab-paclitaxel and gemcitabine showed improved efficacy with acceptable toxicity in this disease setting in first-line and was approved for this indication. The study design allowed patients in standard treatment to receive the combination treatment after first tumour progression.

The proposed study explored the impact of treatment on the QOL scores and compared the times to definitive deterioration of the QOL scores using the validated EORTC QLQ-C30 questionnaire. Efficacy and safety were secondary endpoints and were reported descriptively.

Molecular studies will be performed on blood and tissue samples as avaialble and will be reported separately.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (+ optional for TR) must be given according to ICH/GCP and national/local regulations.
* Patient is at least 18 years of age .
* Unresectable locally advanced or metastatic pancreatic cancer.
* Histologically or cytologically confirmed adenocarcinoma of the pancreas. Islet cell neoplasms are excluded.
* Evaluable or measurable disease, not in a previously irradiated area.
* Life expectancy of at least 12 weeks.
* WHO ECOG performance status ≤ 2
* Adequate organ function.
* Adequate bone marrow, hepatic and renal function. Acceptable coagulation (prothrombin time and partial thromboplastin time within +/- 15% of normal limits).
* No clinically significant abnormalities in urinalysis.
* Effective contraception for both male and female patients if applicable. Women of childbearing potential must have negative blood pregnancy test at screening visit.

Exclusion criteria:

* Prior chemotherapy, radiotherapy, surgery or other investigational therapy for the treatment for metastatic disease. Adjuvant treatment with gemcitabine or 5-FU is allowed provided at least 6 months have elapsed since completion of the last dose.
* Major surgery within 4 weeks of the start of the study.
* Irradiation within 3 weeks prior to study entry.
* Brain metastasis (known or suspected).
* Serious medical risk factors involving any of the major organ systems, including high cardiovascular risk including coronary stenting or myocardial infarction in the last year and psychiatric disorders.
* Historical or active infection with HIV, hepatitis B or C.
* History of connective tissue disorders (eg. lupus, scleroderma, arteritis nodosa, etc).
* History of interstitial lung disease.
* History of peripheral artery disease.
* Previous (within 5 years) or concurrent malignancies at other sites with the exception of surgically cured or adequately treated carcinoma in-situ of the cervix and basal cell carcinoma of the skin.
* Known allergy or any other adverse reaction to any of the drugs or to any related compound.
* Use of Coumadin.
* Organ allografts requiring immunosuppressive therapy.
* Pregnancy or breast-feeding.
* Medical, social or psychological condition which, in the opinion of the investigator, would not permit the patient to complete the study or sign meaningful informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Cutsem, MD, Principal Investigator — UZ Leuven
Locations (18):
- Belgium (18):
  - OLV Ziekenhuis Aalst, Aalst
  - AZ Klina, Brasschaat
  - AZ St Lucas, Bruges
  - ULB Hôpital Erasme, Brussels
  - Cliniques Universitaires St Luc, Brussels
  - CHU de Charleroi, Charleroi
  - UZ Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Heilig Hartziekenhuis Lier, Lier
  - CHC St Joseph, Liège
  - CHR Citadelle, Liège
  - CHU Sart-Tilman, Liège
  - AZ Sint Maarten, Mechelen
  - Clinique St Elisabeth, Namur
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. — http://www.ncbi.nlm.nih.gov/pubmed/8433390
- See also: Quality-of-life (QoL) as a predictive biomarker in patients with advanced pancreatic cancer (APC) receiving chemotherapy: results from a prospective multicenter phase 2 trial. — http://www.ncbi.nlm.nih.gov/pubmed/25436122
- See also: Time until definitive quality of life score deterioration as a means of longitudinal analysis for treatment trials in patients with metastatic pancreatic adenocarcinoma. — http://www.ncbi.nlm.nih.gov/pubmed/20724140
- See also: Pancreatic cancer: optimizing treatment options, new, and emerging targeted therapies. — http://www.ncbi.nlm.nih.gov/pubmed/26185420
- See also: Quality, interpretation and presentation of European Organisation for Research and Treatment of Cancer quality of life questionnaire core 30 data in randomised controlled trials — http://www.ncbi.nlm.nih.gov/pubmed/18599286
- See also: FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer — http://www.ncbi.nlm.nih.gov/pubmed/21561347
- See also: nab-Paclitaxel plus gemcitabine for metastatic pancreatic cancer: long-term survival from a phase III trial. — http://www.ncbi.nlm.nih.gov/pubmed/25638248
- See also: Impact of FOLFIRINOX compared with gemcitabine on quality of life in patients with metastatic pancreatic cancer: results from the PRODIGE 4/ACCORD 11 randomized trial. — http://www.ncbi.nlm.nih.gov/pubmed/23213101
- See also: Minimal important differences for interpreting health-related quality of life scores from the EORTC QLQ-C30 in lung cancer patients participating in randomized controlled trials. — http://www.ncbi.nlm.nih.gov/pubmed/20886240
- See also: Quality of life data as prognostic indicators of survival in cancer patients: an overview of the literature from 1982 to 2008. — http://www.ncbi.nlm.nih.gov/pubmed/20030832
- See also: Impact of the occurrence of a response shift on the determination of the minimal important difference in a health-related quality of life score over time. — http://www.ncbi.nlm.nih.gov/pubmed/27914467
- See also: Baseline quality of life as a prognostic indicator of survival: a meta-analysis of individual patient data from EORTC clinical trials. — http://www.ncbi.nlm.nih.gov/pubmed/19695956
- See also: A global analysis of multitrial data investigating quality of life and symptoms as prognostic factors for survival in different tumor sites. — http://www.ncbi.nlm.nih.gov/pubmed/24127333
- See also: Pancreatic adenocarcinoma. — http://www.ncbi.nlm.nih.gov/pubmed/25207767
- See also: Metastatic Pancreatic Cancer: American Society of Clinical Oncology Clinical Practice Guideline — http://www.ncbi.nlm.nih.gov/pubmed/27247222
- See also: Metastatic Pancreatic Cancer: American Society of Clinical Oncology Clinical Practice Guideline Summary.Metastatic Pancreatic Cancer: American Society of Clinical Oncology Clinical Practice Guideline Summary. — http://www.ncbi.nlm.nih.gov/pubmed/28399388
- See also: Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial. — http://www.ncbi.nlm.nih.gov/pubmed/21969517
- See also: Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. — http://www.ncbi.nlm.nih.gov/pubmed/24131140
- See also: Metastatic Pancreatic Cancer: ASCO Clinical Practice Guideline Update. — http://www.ncbi.nlm.nih.gov/pubmed/29791286
- See also: Joint modeling of longitudinal health-related quality of life data and survival — http://www.ncbi.nlm.nih.gov/pubmed/25311306
- See also: Longitudinal quality of life data: a comparison of continuous and ordinal approaches — http://www.ncbi.nlm.nih.gov/pubmed/24902940
- See also: The role of the FOLFIRINOX regimen for advanced pancreatic cancer — http://www.ncbi.nlm.nih.gov/pubmed/23341367

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred fourty-six patients (pt) were included. First pt enrolled: 08-May-2014. Last pt enrolled: 25-Nov-2015. End of trial notification: 15-May-2018 (last pt last visit) and submitted to ethics committee and competent authorities 10-Jul-2018. Last follow-up (FU) data collected 05-Feb-2019. Cut off date for final data was on 29-Apr-2019.
Groups:
- Arm A (Nab-Paclitaxel + Gemcitabine): Patients were randomised to receive a combination regimen of nab-paclitaxel and gemcitabine.
  Nab-paclitaxel - IV - 125 mg/m2 Schedule: Infusions repeated for three weeks followed by a week of rest (4 week cycles). Nab-paclitaxel infusions were planned every 7 days on the same day of the week; deviations more than 2 days were not allowed.
  Gemcitabine - IV - 1000 mg/m2 Schedule: For patients in Arm A, gemcitabine was given the same day with and following nab-paclitaxel, i.e. once weekly for 3 weeks followed by a week of rest then repeat (4 week cycles). Gemcitabine infusions were planned every 7 days on the same day of the week; deviations more than 2 days were not allowed.
- Arm B (Gemcitabine): Patients were randomised to receive gemcitabine monotherapy.
  Gemcitabine - IV - 1000 mg/m2 Schedule: For patients in Arm B, gemcitabine was given in an initial sequence of seven weeks followed by a week of rest (first cycle is 8 weeks) then every week for three weeks followed by a week of rest (cycle 2 and subsequent cycles are of 4 weeks). Gemcitabine infusions were planned every 7 days on the same day of the week; deviations more than 2 days were not allowed. Patients in Arm B progressing on gemcitabine monotherapy and eligible to receive nab-paclitaxel and gemcitabine were allowed to switch to the combination.
Period: Overall Study
Arm/Group | Arm A (Nab-Paclitaxel + Gemcitabine) | Arm B (Gemcitabine)
Started | 72 | 74
Completed | 72 | 73 (ITT analysis based on treatment assigned at baseline.)
Not Completed | 0 | 1
Not completed — Change of diagnosis/exclusion | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm B (Gemcitabine Monotherapy): Patients were randomised to receive gemcitabine monotherapy.
  Gemcitabine - IV - 1000 mg/m2 Schedule: For patients in Arm B, gemcitabine was given in an initial sequence of seven weeks followed by a week of rest (first cycle is 8 weeks) then every week for three weeks followed by a week of rest (cycle 2 and subsequent cycles are of 4 weeks). Gemcitabine infusions were planned every 7 days on the same day of the week; deviations more than 2 days were not allowed. Patients in Arm B progressing on gemcitabine monotherapy and eligible to receive nab-paclitaxel and gemcitabine were allowed to switch to the combination.
- Total: Total of all reporting groups
Arm/Group | Arm A (Nab-Paclitaxel + Gemcitabine) | Arm B (Gemcitabine Monotherapy) | Total
Number analyzed (Participants) | 72 | 74 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 37 | 76
  >=65 years | 33 | 37 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 41 | 42 | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ECOG performance status [Count of Participants; unit: Participants] — WHO EGOG performance status (PS) scale 0 Able to carry out all normal activity without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out light work
  2. Ambulatory and capable of all self-care but unable to carry out any work; up and about more than 50% of waking hours.
  3. Capable of only limited self-care; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair
  Participants
    0 | 27 | 23 | 50
    1 | 42 | 49 | 91
    2 | 3 | 2 | 5
Site of pancreatic tumor [Count of Participants; unit: Participants]
  Head | 16 | 19 | 35
  Body | 37 | 34 | 71
  Tail | 19 | 21 | 40
Locally advanced / metastatic [Count of Participants; unit: Participants]
  Locally advanced | 10 | 11 | 21
  Metastatic | 62 | 63 | 125
Adjuvant treatment prior to inclusion [Count of Participants; unit: Participants]
  Yes | 5 | 6 | 11
  No | 67 | 68 | 135

OUTCOME MEASURES:

1. Primary Outcome: Deterioration-free Survival Rate of the QOL Global Health Status at 3, 6 and 12 Months (Mos)
Description: The QOL global health status (GHS) is a functional parameter derived from the EORTC QLQ - C30 questionnaire, based on questions 29 "How would you rate your overall health during the past week?" and 30 "How would you rate your overall quality of life during the past week?". Transformed scores range from 0 to 100% with higher scores representing better outcomes. The deterioration free survival rate at 3 mos is defined as the Kaplan-Meier estimate of the probability of being alive and free of deterioration of the QOL score at 3 mos. The definitive deterioration of the QOL score is a decrease of at least 10 points (minimal clinical important difference) as compared to baseline, with no further improvement of more than 10 points as compared to the score qualifying the deterioration or with no data after deterioration. Death was also considered as an event if the patient did not experience deterioration before death. Patients without event were censored at the time of last follow-up.
Time Frame: From date of randomisation to 3, 6 and 12 months respectively
Population: ITT analysis based on the treatment groups randomized at baseline. Pts in Arm B were allowed to switch to the combination treatment after the initial progression but were considered solely in Arm B for this ITT analysis, as per protocol. Subset analyses of combination data in treatment switchers will be published in a peer reviewed journal.
Measure: Number; unit: percentage of participants
Groups:
- Arm B (Gemcitabine): Patients were randomised to receive gemcitabine monotherapy.
  Gemcitabine - IV - 1000 mg/m2 Schedule: For patients in Arm B, gemcitabine was given in an initial sequence of seven weeks followed by a week of rest (first cycle is 8 weeks) then every week for three weeks followed by a week of rest (cycle 2 and subsequent cycles are of 4 weeks). Gemcitabine infusions were planned every 7 days on the same day of the week; deviations more than 2 days were not allowed. Patients in Arm B progressing on gemcitabine monotherapy and eligible to receive nab-paclitaxel and gemcitabine were allowed to switch to the combination (N=37).
Arm/Group | Arm A (Nab-Paclitaxel + Gemcitabine) | Arm B (Gemcitabine)
Number analyzed (Participants) | 72 | 73
percentage of participants
  Rate at 3 months (percentage) | 89 | 73
  Rate at 6 months (percentage) | 74 | 59
  Rate at 12 months (percentage) | 40 | 35

2. Primary Outcome: QOL Global Health Status Deterioration-free Median Survival
Description: The deterioration-free survival is defined as the Kaplan-Meier estimate of median survival time to definitive deterioration of the QOL score or death. See primary outcome 1 for scale description. The definitive deterioration of the QOL score is a decrease of at least 10 points (minimal clinical important difference) as compared to the baseline score, with no further improvement of more than 10 points as compared to the score qualifying the deterioration or with no data after the deterioration was observed. Death was also considered as an event if the patient did not experience deterioration before death. Patients without event were censored at the time of last follow-up.
Time Frame: From date of randomisation to end of follow up (max 3 years after database lock when applicable).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm A (Nab-Paclitaxel +Gemcitabine): Patients were randomised to receive a combination regimen of nab-paclitaxel and gemcitabine.
  Nab-paclitaxel - IV - 125 mg/m2 Schedule: Infusions repeated for three weeks followed by a week of rest (4 week cycles). Nab-paclitaxel infusions were planned every 7 days on the same day of the week; deviations more than 2 days were not allowed.
  Gemcitabine - IV - 1000 mg/m2 Schedule: For patients in Arm A, gemcitabine was given the same day with and following nab-paclitaxel, i.e. once weekly for 3 weeks followed by a week of rest then repeat (4 week cycles). Gemcitabine infusions were planned every 7 days on the same day of the week; deviations more than 2 days were not allowed.
Arm/Group | Arm A (Nab-Paclitaxel +Gemcitabine) | Arm B (Gemcitabine)
Number analyzed (Participants) | 72 | 73
Months | 10.04 [7.16 to 12.02] | 8.02 [5.49 to 11.37]

3. Secondary Outcome: Overall Response
Description: Tumour response was assessed locally based on radiological assessments (CT/MRI) of target and nontarget lesions and considering the occurrence of new lesions, as per RECIST criteria. Tumour response was defined at each evaluation as complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD). Best response during treatment was selected for each patient. Overall response (OR) is defined as the best tumor response on treatment for each patient. Responders were considered CR + PR. Some patients were not evaluable for response (no scans available). Overall response rates (ORR) were calculated based on the ITT set.
Time Frame: Measured during treatment and FU, from signature of informed consent to progression (variable for each patient), for a max of 3 years from database lock (when applicable).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Nab-Paclitaxel + Gemcitabine) | Arm B (Gemcitabine)
Number analyzed (Participants) | 72 | 73
Participants
  CR or PR | 31 | 16
  SD or PD | 39 | 53
  Not evaluable | 2 | 4

4. Secondary Outcome: Duration of Response (in Responders)
Description: Duration of response was calculated from the date of first documented response to the date of progression (including SD after PR) or date of start of new treatment in not progressed, when available. In 2 patients with CR, periods of PR are included. For those not documented as progressed before death, an unknown duration was kept and considered missing data.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Nab-Paclitaxel + Gemcitabine) | Arm B (Gemcitabine)
Number analyzed (Participants) | 72 | 73
Months | 6.3 [1.92 to 35] | 7.4 [1.5 to 20]

5. Secondary Outcome: Disease Control
Description: Tumour response was assessed locally based on radiological assessments (CT/MRI) of target and nontarget lesions and considering the occurrence of new lesions, as per RECIST criteria. Tumour response was defined at each evaluation as complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD). Best response during treatment was selected for each patient. Overall response is defined as the best tumor response on treatment for each patient. Disease control is defined as a best response on treatment of either CR, PR or SD (CR + PR + SD). Some patients were not evaluable for response (no scans available). Overall response rates were calculated based on the ITT set.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Nab-Paclitaxel + Gemcitabine): Patients were randomised to receive a combination regimen of nab-paclitaxel and gemcitabine.
  Nab-paclitaxel) - IV - 125 mg/m2 Schedule: Infusions repeated for three weeks followed by a week of rest (4 week cycles). Nab-paclitaxel infusions were planned every 7 days on the same day of the week; deviations more than 2 days were not allowed.
  Gemcitabine - IV - 1000 mg/m2 Schedule: For patients in Arm A, gemcitabine was given the same day with and following nab-paclitaxel, i.e. once weekly for 3 weeks followed by a week of rest then repeat (4 week cycles). Gemcitabine infusions were planned every 7 days on the same day of the week; deviations more than 2 days were not allowed.
Arm/Group | Arm A (Nab-Paclitaxel + Gemcitabine) | Arm B (Gemcitabine)
Number analyzed (Participants) | 72 | 73
Participants
  CR + PR + SD | 58 | 60
  PD | 12 | 9
  Not evaluable | 2 | 4

6. Secondary Outcome: Progression Free Survival
Description: Progression free survival time was considered from start of treatment until the first observation of disease progression or death from any cause, whichever occurred first. All patients (ITT).
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Nab-Paclitaxel + Gemcitabine) | Arm B (Gemcitabine)
Number analyzed (Participants) | 72 | 73
Months | 7.01 [5.45 to 8.05] | 5.06 [3.52 to 7.00]

7. Secondary Outcome: Overall Survival
Description: Overall survival was considered from start of treatment to death. All patients (ITT)
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Nab-Paclitaxel + Gemcitabine) | Arm B (Gemcitabine)
Number analyzed (Participants) | 72 | 73
Months | 10.94 [8.97 to 15.18] | 11.73 [8.74 to 13.44]

8. Secondary Outcome: Laboratory Safety Assessment
Description: Severe laboratory abnormalities (hematology and biochemistry grade 3 and higher). Worst grade per patient. All patients treated (Safety set).
Time Frame: Measured during treatment, from signature of informed consent to end of treatment, plus 30 days mandatory safety follow-up period. Duration of treatment was variable for each patient.
Population: All pts treated (safety set). Analysis based on the treatment groups randomized at baseline. Pts in Arm B were allowed to switch to the combination treatment after the initial progression but were considered solely in Arm B for this ITT analysis, as per protocol. Subset analyses in treatment switchers will be published in a peer reviewed journal.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Nab-Paclitaxel + Gemcitabine) | Arm B (Gemcitabine)
Number analyzed (Participants) | 72 | 74
Participants
  Hemoglobin decreased | 10 | 8
  Neutrophils decreased | 31 | 31
  White blood cell count decreased | 22 | 11
  Platelet count decreased | 12 | 11
  Hyperglycemia | 6 | 10
  Serum creatinine increased | 0 | 2
  Bilirubin increased | 3 | 8
  ALT increased | 13 | 8
  AST increased | 7 | 8
  ALP increased | 9 | 11
  Albumin decreased | 4 | 4
  Magnesium decreased | 4 | 9
  Sodium decreased | 8 | 13
  Potassium decreased | 8 | 6
  Potassium increased | 1 | 0
  Calcium decreased | 3 | 2

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAE) and adverse events (AE) occurring from the signature of informed consent to the end of treatment visit plus 30 days. Pts in Arm B were allowed to switch to the combination treatment after the initial progression. This ITT analysis reports all AEs for the whole duration of treatment and mandatory safety FU, per arm as randomized at baseline, as per protocol. Subset analyses of combination data in treatment switchers will be published in a peer reviewed journal.
Description: All SAEs occurring between the signature of informed consent and the end of treatment visit + 30 days are listed.
  Severe adverse events (grade 3-5, worst grade per patient) are listed in the section " Other Adverse Events" , SAEs are included.
  A summary of the severe laboratory abnormalities is provided in section "End points".
Groups:
- Arm A (Nab-Paclitaxel + Gemcitabine): Nab-paclitaxel - IV - 125 mg/m2 - 3xq4wks Gemcitabine - IV - 1000 mg/m2 - 3xq4wks
- Arm B (Gemcitabine): Gemcitabine - IV - 1000 mg/m2 - 3xq4wks
Arm/Group | Arm A (Nab-Paclitaxel + Gemcitabine) | Arm B (Gemcitabine)
All-Cause Mortality (participants affected / at risk) | 5/72 | 11/74
Serious Adverse Events (participants affected / at risk) | 50/72 | 48/74
Other Adverse Events (participants affected / at risk) | 72/72 | 74/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Nab-Paclitaxel + Gemcitabine) (N=72) | Arm B (Gemcitabine) (N=74)
Thromboembolic event (Vascular disorders) | 3 (5) | 3 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 5 (5)
Fever (General disorders) | 9 (10) | 9 (10)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 3 (3) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Alteration of general condition (General disorders) | 0 (0) | 1 (1)
Drug misuse (General disorders) | 0 (0) | 1 (1)
Generalized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Galbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemolytic Uremic Syndrome (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal and galbladder obstruction on stent (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastro-enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sigmoiditis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic duct stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (4)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 3 (4)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (3)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Jaundice (Hepatobiliary disorders) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 3 (4)
Major denutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (2) | 0 (0)
Biliary tract infection (Infections and infestations) | 3 (3) | 3 (3)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 7 (9) | 2 (2)
Infectious syndrome (Infections and infestations) | 1 (1) | 0 (0)
Infectious exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Septic thromboflebitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Nab-Paclitaxel + Gemcitabine) (N=72) | Arm B (Gemcitabine) (N=74)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 8 (12) | 7 (11)
Thromboembolic event (Vascular disorders) | 5 (6) | 6 (8)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 16 (26) | 21 (38)
Fever (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
General status altteration (General disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 1 (2) | 5 (5)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (2) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 7 (9) | 11 (18)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (6) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 2 (3) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 8 (9)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colinic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 6 (6)
Obstruction gastric (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intrapancreatic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernia inguinalis with obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Small intestinal onstruction (Gastrointestinal disorders) | 2 (2) | 2 (3)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper GI haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 4 (4)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3)
Bile duct stenosis (Hepatobiliary disorders) | 2 (2) | 6 (6)
Cholecystitis (Gastrointestinal disorders) | 1 (1) | 4 (6)
Galbladder obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 2 (3)
Dilated bile ducts (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Hepatobiliary disorders) | 1 (2) | 0 (0)
Pain in extremity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (8) | 14 (18)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Abdominal infection (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Galbladder infection (Infections and infestations) | 1 (2) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (2) | 1 (2)
Lung infection (Infections and infestations) | 6 (7) | 3 (3)
Infection without neutropenia NOS (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
Quality of life endpoints are sensitive to confounding factors such as age, intercurrent disease, time from last completed questionnaire to the last follow-up or death. Tumour response and AE relationship to treatment were locally adressed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT02106884/Prot_SAP_000.pdf